CLINICAL TRIAL: NCT03328507
Title: A Pilot Evaluation of BLI4900 Bowel Preparation in Adult Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BLI4900-201
Record Dates: First submitted 2017-10-30; First posted 2017-11-01 (Actual); Results first posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-09

CONDITIONS: Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BLI4900 (Experimental): BLI4900 Bowel Preparation
  Interventions: Drug: BLI4900
- PEG Control (Active Comparator): Polyethylene glycol-based bowel preparation
  Interventions: Drug: PEG Control

INTERVENTIONS:
Drug: BLI4900 — BLI4900 Bowel Preparation
  Arms: BLI4900
Drug: PEG Control — Polyethylene glycol-based bowel preparation
  Arms: PEG Control

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of BLI4900 as a bowel preparation prior to colonoscopy in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients who are undergoing colonoscopy for a routinely accepted indication.
* 18 to 85 years of age (inclusive).
* If female, and of child-bearing potential, is using an acceptable form of birth control (hormonal birth control, IUD, double-barrier method, depot contraceptive, abstinent, or vasectomized spouse).
* Negative urine pregnancy test at screening, if applicable.
* In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study.

Exclusion Criteria:

* Subjects with known or suspected ileus, severe ulcerative colitis, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis or megacolon.
* Subjects with ongoing severe, acute inflammatory bowel disease.
* Subjects who had previous significant gastrointestinal surgeries.
* Subjects with uncontrolled pre-existing electrolyte abnormalities, or those with clinically significant electrolyte abnormalities based on Visit 1 laboratory results.
* Subjects with uncontrolled hypertension (systolic blood pressure > 170 mmHg and diastolic blood pressure > 100 mmHg).
* Subjects with severe renal insufficiency (GFR < 30 mL/min/1.73m2).
* Subjects with known severe hepatic insufficiency (Child Pugh C).
* Subjects with cardiac insufficiency (NYHA Functional Classifications 3 or 4).
* Subjects undergoing insulin therapy for any indication.
* Subjects with impaired consciousness that predisposes them to pulmonary aspiration.
* Subjects undergoing colonoscopy for foreign body removal and/or decompression.
* Subjects who are pregnant or lactating, or intending to become pregnant during the study.
* Subjects of childbearing potential who refuse a pregnancy test.
* Subjects allergic to any preparation components.
* Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures.
* Subjects who have participated in an investigational surgical, drug, or device study within the past 30 days.
* Subjects who withdraw consent before completion of Visit 1 procedures.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, MPH, Study Director — Braintree Laboratories, Inc.
Locations (4):
- United States (4):
  - Braintree Research Site 1, Anaheim, California
  - Braintree Research Site 3, Chula Vista, California
  - Braintree Research Site 4, San Diego, California
  - Braintree Clinical Research Site 2, Ogden, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wiener G, Winkle P, McGowan JD, Cleveland MV, Di Palma JA. A Phase 2 evaluation of a new flavored peg and sulfate solution compared to an over-the-counter laxative, peg and sports drink bowel preparation combination. BMC Gastroenterol. 2023 Dec 11;23(1):433. doi: 10.1186/s12876-023-03069-8. PMID 38082231

RESULTS

PARTICIPANT FLOW:
Groups:
- BLI4900-3: Formulation 3
- BLI4900-5: Formulation 5
- BLI4900-6: Formulation 6
- PEG-SD: Polyethylene glycol 3350 mixed with sports drink (plus bisacodyl)
Period: Overall Study
Arm/Group | BLI4900-3 | BLI4900-5 | BLI4900-6 | PEG-SD
Started | 21 | 40 | 41 | 19
Completed | 21 | 40 | 40 | 19
Not Completed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BLI4900-3 | BLI4900-5 | BLI4900-6 | PEG-SD | Total
Number analyzed (Participants) | 21 | 40 | 40 | 19 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (11.1) | 54.5 (11.5) | 58.7 (10.2) | 49.7 (15.7) | 55.2 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 20 | 24 | 12 | 66
  Male | 11 | 20 | 16 | 7 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 15 | 7 | 28
  Not Hispanic or Latino | 16 | 39 | 25 | 12 | 92
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 0 | 6 | 4 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2 | 0 | 4
  Black or African American | 0 | 0 | 3 | 1 | 4
  White | 17 | 38 | 29 | 14 | 98
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 40 | 40 | 19 | 120

OUTCOME MEASURES:

1. Primary Outcome: % of Subjects With Successful Bowel Preparation
Description: % of subjects with successful bowel preparation rated by blinded colonoscopist on a 4 point scale (1=poor to 4 = excellent)
Time Frame: Day of colonoscopy
Measure: Count of Participants; unit: Participants
Arm/Group | BLI4900-3 | BLI4900-5 | BLI4900-6 | PEG-SD
Number analyzed (Participants) | 21 | 40 | 40 | 19
Participants | 17 | 37 | 37 | 16

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | BLI4900-3 | BLI4900-5 | BLI4900-6 | PEG-SD
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/40 | 0/41 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/40 | 0/41 | 1/19
Other Adverse Events (participants affected / at risk) | 13/21 | 31/40 | 13/41 | 14/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BLI4900-3 (N=21) | BLI4900-5 (N=40) | BLI4900-6 (N=41) | PEG-SD (N=19)
diverticulitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BLI4900-3 (N=21) | BLI4900-5 (N=40) | BLI4900-6 (N=41) | PEG-SD (N=19)
abdominal distension (Gastrointestinal disorders) | 11 | 26 | 8 | 10
abdominal pain upper (Gastrointestinal disorders) | 7 | 17 | 6 | 5
nausea (Gastrointestinal disorders) | 7 | 19 | 5 | 7
vomiting (Gastrointestinal disorders) | 3 | 2 | 3 | 1
hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
headache (Nervous system disorders) | 2 | 0 | 0 | 0
migraine (Nervous system disorders) | 1 | 0 | 0 | 0
orthostatic hypotension (Vascular disorders) | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sole disclosure restriction which sponsor imposes on the PI is a sixty (60) day limited restriction in order to the protect potentially proprietary information which may be patentable.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT03328507/Prot_SAP_000.pdf